CLINICAL TRIAL: NCT06466642
Title: Building Resources to Achieve Improvement in Neurocognition (B.R.A.I.N) in People Living With HIV
Brief Title: B.R.A.I.N in People Living With HIV Study
Acronym: BRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, KevinThomas, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 045-2022
Record Dates: First submitted 2024-05-22; First posted 2024-06-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: HIV-associated Neurocognitive Disorders
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Recruited participants will first be screened for eligibility and required to provide informed consent. After the baseline assessment, participants will be randomized into one of two study arms: an active experimental group receiving CR (CogSMART and BrainHQ©) or an attention-matched control group. Measures, both subjective and objective, will evaluate participants' cognition, behavior, and functional abilities. Exit focus groups will gather participant feedback. The study aims to inform a larger RCT to enhance cognitive functioning and well-being among PWH in South Africa.
Who Masked: Outcomes Assessor
Masking Description: Randomization to study arm. Participants will be randomized into one of two study arms after the baseline assessment: an active experimental group receiving the CR, or an attention-matched control group. Because our sample size (N=43) is smaller than 100, investigators will use block randomization to assign participant numbers equally across each arm. To prevent the executer (the neuropsychology technician) from predicting the next assignment, they will be kept ignorant of the block size. Concealing the allocation sequence from those assigning participants, will prevent selection bias. Allocation numbers will be placed in individually sealed brown envelopes by the project manager prior to study commencement.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined CogSMART and BrainHQ intervention group (Experimental): Intervention: The experimental condition in this trial is a combination of CogSMART and BrainHQ. This integrated intervention helps individuals with cognitive impairment improve daily activities and achieve goals. CogSMART, a compensatory cognitive remediation (C-CR) program, employs techniques to enhance prospective memory, attention, learning/memory, and executive functioning. BrainHQ, a restorative cognitive remediation (R-CR) program, provides game-like modules targeting memory, attention, and executive functions. Together, they offer a comprehensive approach, combining C-CR with R-CR to reduce impairment and enhance problem-solving skills.
  Interventions: Behavioral: Combined Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) and BrainHQ©
- Attention-matched Combined CogSMART and BrainHQ Control group (No Intervention): This control-matched approach to the CogSMART group, currently utilized in Dr. Twamley's studies, has been well received by participants, with no significant increase in dropout rates. Additionally, control participants will receive the BrainHQ component, involving Internet Navigation Training previously employed by Dr. Vance consisting of 20 sessions lasting 30 minutes each aimed to provide no therapeutic benefit.

INTERVENTIONS:
Behavioral: Combined Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) and BrainHQ© — The intervention combines Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) and BrainHQ. This integrated program helps individuals with cognitive impairment improve daily activities and achieve work, social, and daily living goals. CogSMART uses compensatory techniques to enhance prospective memory (remembering to do things), attention, learning/memory, and executive functioning (problem-solving, planning, organization, and cognitive flexibility). BrainHQ complements CogSMART with stimulating, game-like modules focusing on memory, attention, and executive functions. Together, they provide a comprehensive therapeutic tool to support cognitive impairment treatments and can also be used as a brain-training tool to prevent memory loss and maintain cognitive abilities.
  Arms: Combined CogSMART and BrainHQ intervention group

SUMMARY:
People living with HIV (PLWH) often have memory and thinking problems, which can range from mild to severe. These problems, which are called neurocognitive impairment (NCI), can appear even when PLWH are taking medicine to manage their HIV.

PLWH who are experiencing NCI can have difficulties managing everyday activities. For instance, they might not remember to take their medicine on time, they might struggle to manage their money properly, and they might even be at a higher risk of passing HIV on to other. Ultimately, PLWH who are experiencing NCI might not enjoy life as much as others do.

Currently, there are no specific medicines designed to treat NCI in PLWH. There are, however, some useful memory and thinking strategies that can help improve cognitive abilities. These strategies are called cognitive remediation (CR).

In South Africa, there are many PLWH. Unfortunately, the country does not have clear plans for identifying and managing NCI in PLWH. It's difficult to use CR in South Africa because of cultural differences between where the strategies were developed and the patients who might need to use it, limited healthcare resources, and HIV clinics not having enough information about NCI.

There are, however, some promising ways to deal with these issues. For example, it can be helpful to involve regular counselors and to use simple tests on mobile phones to find people who need assistance. With some effort and creativity, investigators can improve the situation and help PLWH lead better lives.

The proposed study is a unique opportunity to find new ways to help PLWH and others with brain-related diseases who might be experiencing NCI. Investigators want to explore ways to use cognitive exercises to improve thinking abilities. This study will be the first of its kind because investigators will adapt these exercises to fit the cultures and languages of South Africa, where many people are affected by HIV and NCI.

By doing this research, investigators hope to make important progress in addressing NCI in HIV and similar conditions. Investigators will learn how to make these cognitive exercises work best in South Africa's public clinics, and this knowledge can help people with NCI live better lives. Our goal is to improve healthcare not only in South Africa but also in other parts of the world that might be facing similar challenges with improving the lives of PLWH.

DETAILED DESCRIPTION:
Neurocognitive Impairment (NCI) is a condition where HIV infection affects the brain, leading to problems with memory, thinking, and other cognitive functions. It is a common issue among people living with HIV, even those who are receiving antiretroviral therapy (ART) to control the virus. The exact reasons why NCI occurs in HIV are not fully understood, but it is likely influenced by several factors, including direct HIV-related processes in the central nervous system and other contributing elements like stress.

NCI can range from mild cognitive deficits to more severe impairments that impact daily functioning and quality of life. People experiencing NCI may find it challenging to remember things, concentrate, make decisions, and perform tasks they once managed easily. This condition can also affect their adherence to HIV treatment, which is crucial for managing the infection effectively.

In South Africa, where HIV prevalence is high, NCI poses a significant concern. Despite its prevalence, there are no established protocols for the routine screening and management of NCI in HIV clinics. This lack of systematic approach hinders early identification and appropriate intervention for affected individuals.

The consequences of NCI in HIV are not just medical; they extend to functional and public health aspects as well. For instance, impaired cognitive abilities can hinder a person's ability to adhere to their medication schedule, leading to treatment challenges and potential disease progression. Additionally, NCI can hinder daily activities and job performance, affecting overall productivity and livelihood. Furthermore, those with cognitive impairments may be at a higher risk of transmitting HIV to others, as they might struggle with understanding and adhering to preventive measures.

Currently, there are no specific pharmacological treatments available to directly address NCI in HIV. However, cognitive remediation (CR) strategies have shown promise in managing and improving cognitive abilities in this population. CR involves structured activities and exercises designed to enhance memory, attention, problem-solving, and other cognitive functions. While more research is needed, CR holds potential for improving the quality of life for individuals living with HIV and NCI.

Implementing CR interventions in South Africa faces several challenges. The country's cultural diversity calls for approaches that are sensitive and adaptable to different communities. Moreover, limited healthcare resources and the lack of awareness and guidelines for NCI in HIV clinics add further complexity to the situation.

One promising approach involves task-shifting strategies, which involve the participation of lay counselors in the delivery of CR interventions. This can help address resource constraints while potentially reaching more affected individuals. Additionally, utilizing mobile health screening tests can aid in identifying people with NCI, especially in remote or underserved areas.

The proposed study provides a unique opportunity to establish an entirely new therapeutic approach on the African continent for treating neurocognitive impairment (NCI) in people living with HIV (PWH) and patients with other brain-involved diseases. Additionally, it aims to explore barriers to the utility and future implementation of cognitive remediation (CR) in public clinics.

This study will be the first of its kind in several ways: (1) It will culturally and linguistically adapt a CR program specifically for HIV-associated NCI in a low- and middle-income setting with high rates of HIV and NCI; (2) It will assess the usability and acceptability of the CR intervention by both key stakeholders, such as the Department of Health, and PWH in South Africa; (3) It will combine evidence-based restorative and compensatory cognitive remediation strategies and evaluate which components are most acceptable and feasible to implement in the South African context.

By undertaking this groundbreaking research, investigators aim to make significant strides in addressing NCI in HIV and potentially extend the benefits to other brain-involved conditions. The study's outcomes will provide valuable insights into the implementation of CR in the country's public clinics and pave the way for more effective and culturally appropriate interventions for improving cognitive function in those affected by HIV-associated NCI and other related diseases. Through this collaborative effort, investigators hope to improve the lives of individuals living with NCI and contribute to the advancement of healthcare in South Africa and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 50 years;
* ≥ 8 years of schooling;
* Fluent Xhosa speaking;
* HIV-positive;
* on Antiretroviral therapy (ART);
* ability to sign informed consent;
* willing to attend: (a) two NP testing sessions, (b) a minimum of 10 hours (twenty 30-minute sessions) of R-CR sessions, and (c) 10 CogSMART sessions over a period of five weeks; and
* meeting the criteria for NCI (as described further in document).

Exclusion Criteria:

* Participants with significant neuro-medical comorbidities (e.g., schizophrenia, epilepsy, bipolar disorder, multiple sclerosis, intellectual disability) necessitate exclusion. These comorbidities will be assessed for during screening.
* Other conditions (e.g., legally blind or deaf, currently undergoing radiation or chemotherapy, a history of brain trauma with a loss of consciousness greater than 30 minutes) that could impact cognitive functioning, testing or consistent study participation over 7 weeks necessitate exclusion; again, this information is conferred in the screen.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessment: Learning and Memory (1) | 10 weeks
  Hopkins Verbal Learning Test Total Recall: Measures verbal learning and memory. Scores range from 0 to 30, with higher scores indicating better memory retention. Task done over 20 minutes.
Neuropsychological assessment: Learning and Memory (2) | 10 weeks
  Hopkins Verbal Learning Test Delayed Recall: Assesses delayed verbal recall. Scores range from 0 to 12, reflecting the ability to retain information. Task done over 20 minutes.
Neuropsychological assessment: Learning and Memory (3) | 10 weeks
  Wechsler Adult Intelligence Scale-III Digit Span Total: Evaluates auditory attention and working memory. Scores range from 0 to 16, with higher scores indicating better performance in recalling sequences of digits.
Neuropsychological assessment: Processing Speed (1) | 10 weeks
  Wechsler Adult Intelligence Scale-III Symbol Search Total: Assesses processing speed and attention. Scores range from 0 to 60, with higher scores indicating better performance in quickly identifying matching symbols. This task is done in 120 seconds.
Neuropsychological assessment: Processing Speed (2) | 10 weeks
  Wechsler Adult Intelligence Scale-III Coding Total: Evaluates processing speed, attention, and visual-motor coordination. Scores range from 3 to 70, with higher scores indicating faster completion of the coding task.
Neuropsychological assessment: Processing Speed (3) | 10 weeks
  Trail Making Test Part A Time: Evaluates processing speed, visual attention, and task-switching ability. Scores range from 0 to 158 seconds, with lower times indicating better performance in processing speed, visual attention and task-switching ability, as they reflect faster task completion without errors
Neuropsychological assessment: Processing Speed (4) | 10 weeks
  Trail Making Test Part A Time (Extended): This extended version of the Trail Making Test Part A measures processing speed, with scores ranging from 0 to 300 seconds. Lower times indicate better performance, as they reflect quicker task completion without errors.
Neuropsychological assessment: Executive Functioning (1) | 10 weeks
  Semantic Fluency Animals Correct: Assesses language and executive function over 60 seconds. Scores range from 0 to 22, with higher scores indicating greater fluency.
Neuropsychological assessment: Executive Functioning (2) | 10 weeks
  Semantic Fluency Fruit/Vegetable Correct: Evaluates semantic fluency for fruits and vegetables over 60 seconds. Scores can range from 0 to 22, reflecting the participant's ability to generate words within this category.
Neuropsychological assessment: Executive Functioning (3) | 10 weeks
  Grooved Pegboard Test Dominant Hand Time: This test evaluates fine motor skills and coordination in the dominant hand. Scores range from 0 to 160 seconds, with lower times indicating better manual dexterity and motor coordination.
Neuropsychological assessment: Executive Functioning (4) | 10 weeks
  Grooved Pegboard Test Non-Dominant Hand Time: Assesses fine motor skills and coordination for the non-dominant hand. Scores range from 60 to 300 seconds, with lower times indicating better manual dexterity and motor coordination.

SECONDARY OUTCOMES:
HIV outcomes: ART Adherence (Dried Blood Spot Analysis) (1) | 5 weeks
  * Assessment Used: Measurement of Tenofovir Diphosphate Levels
  * Units of Measure: Concentration (ng/mL)
  * Minimum: 10 ng/mL
  * Maximum: 2000 ng/mL
  * Description: Dried blood spots will be collected and analyzed to measure tenofovir diphosphate levels as a marker of ART adherence. Higher concentrations of tenofovir diphosphate indicate better adherence to antiretroviral therapy.
HIV outcomes: Systemic Inflammation (Dried Blood Spot Analysis) (2) | 5 weeks
  * Assessment Used: Measurement of Interleukin-6 Levels
  * Units of Measure: Concentration (pg/mL)
  * Minimum: 0.5 pg/mL
  * Maximum: 500 pg/mL
  * Description: Dried blood spots will be analyzed to measure interleukin-6, a pro-inflammatory cytokine linked to neurocognitive impairment. Higher concentrations of interleukin-6 indicate greater levels of systemic inflammation.
HIV outcomes: Self-Reported ART Adherence (3) | 5 weeks
  * Assessment Used: Three-item Self-Report Medication Adherence Scale
  * Units of Measure: Adherence score (0-3)
  * Minimum: 0
  * Maximum: 3
  * Description: Participants will self-report their ART adherence using a three-item scale, providing a subjective measure of adherence. Higher scores indicate better self-reported adherence to antiretroviral therapy.

OTHER OUTCOMES:
Other Study Measures: Mood Disorders (1) | 5 weeks
  Center for Epidemiologic Studies Depression Scale: Measures symptoms of depression. Scores; minimum 0, maximum 60. Higher scores indicate greater severity.
Other Study Measures: Mood Disorders (2) | 5 weeks
  Patient Health Questionnaire-2: Measures frequency of depressed mood and anhedonia over the past 5 weeks. Scores; minimum 0, maximum 6. Higher scores indicate greater severity.
Other Study Measures: Post-Traumatic Stress | 5 weeks
  Primary Care Post Traumatic Stress Disorder Screen: Measures symptoms of post-traumatic stress disorder. Scores; minimum 0, maximum 6. Higher scores indicate greater severity.
Other Study Measures: Physical Functioning | 5 weeks
  World Health Organization Disability Assessment Schedule: Measures general health and disability. Scores; minimum 0, maximum 100. Higher scores indicate greater disability.
Other Study Measures: Disease-Specific Quality of Life | 5 weeks
  Ability to Perform Social Roles and Activities: Measures ability to perform social roles and activities. Scores; minimum 0, maximum 100. Higher scores indicate better social functioning.
Other Study Measures: Adherence | 5 weeks
  Adherence Questionnaire: Measures adherence to treatment or prescribed interventions. Scores; minimum 0, maximum 100. Higher scores indicate better adherence.
Other Study Measures: Communication skills | 5 weeks
  World Health Organization Disability Assessment Schedule: Measures communication difficulties. Scores; minimum 0, maximum 100. Higher scores indicate more disability.
Other Study Measures: Anxiety | 5 weeks
  Generalized Anxiety Disorder Scale: Measures severity of generalized anxiety disorder. Scores; minimum 0, maximum 21. Higher scores indicate more severe anxiety.
Other Study Measures: Neurobehavioral Symptom | 5 weeks
  Neurobehavioral Symptom Inventory: Measures severity of neurobehavioral symptoms such as headache, dizziness, and irritability. Scores; minimum 0, maximum 88. Higher scores indicate more severe symptoms.
Other Study Measures: Quality of Life | 5 weeks
  Patient-Reported Outcomes Measurement Information System T-score: Measures general health and well-being. Higher scores indicate better quality of life.
Other Study Measures: Psychological Distress | 5 weeks
  Stress and Anxiety Symptom Scale - Bothered: Measures level of psychological distress and how bothered the individual feels, scores; minimum 0, maximum 100. Higher scores indicate more distress.
Other Measures: Cognitive Skills: Applied Cognition General Concerns Scale (1) | 5 weeks
  Measures general concerns about cognitive functioning, including memory, attention, and executive function. Scores: maximum 0, minimum 36. Scores indicate the level of concern an individual has about their cognitive abilities, with higher scores suggesting more concerns.
Other Measures: Cognitive Skills: Applied Cognition Executive Functions Total Scale (2) | 5 weeks
  Measures executive functions, including planning, problem-solving, and cognitive flexibility. Scores minimum 0, maximum 40. Scores indicate the degree of impairment in executive functions, with higher scores indicating more severe impairment.
Other Measures: Cognitive Skills: Cognitive Problems and Strategies Assessment Strategies Total Scale (3) | 5 weeks
  The Cognitive Problems and Strategies Assessment Total Scale evaluates memory-related cognitive issues and the effectiveness of coping strategies. It measures the severity of memory problems and how frequently individuals use cognitive strategies to manage them, scoring; a minimum of 0, and a maximum of 90. Higher scores indicate more severe cognitive issues and more frequent use of coping strategies.
Other Measures: Cognitive Skills: Patient's Assessment of Own Functioning High Frequency Total Scale (4) | 5 weeks
  Measures high-frequency cognitive functioning, including attention, memory, and executive function. Scores; minimum 0, maximum 55. Scores indicate the level of impairment in high-frequency cognitive tasks, with higher scores suggesting more impairment.
Other Measures: Cognitive Skills: Patient's Assessment of Own Functioning Memory Total Scale (5) | 5 weeks
  Measures memory-related cognitive functioning, including recall and recognition. Scores; minimum 0, maximum 60. Scores indicate the level of impairment in memory-related cognitive tasks, with higher scores indicating more severe impairment in memory function.
Other Study Measures: Exit Interviews | 10 weeks
  The assessment used is a structured exit interview questionnaire, to explore participants' subjective experiences and perceived benefits of the intervention. The units of measure will be qualitative themes and sub-themes identified from participant responses. A thematic analysis will be conducted to identify common themes.
Other Study Measures: Focus Group Discussion | 10 weeks
  The assessment will utilize a structured focus group discussion guide to explore the collective views and experiences of the participants regarding the intervention. The units of measure will be qualitative themes and sub-themes identified from the group discussion. Thematic analysis will be conducted to identify common themes.

CONTACTS AND LOCATIONS:
Overall Officials: Hetta Gouse, PhD, Principal Investigator — University of Cape Town; John Joska, PhD, Principal Investigator — University of Cape Town
Locations (3):
- South Africa (3):
  - Michael Mapongwana Community Health Clinic, Cape Town, Western Cape
  - TB HIV Care, Cape Town, Western Cape
  - Nolungile Community Clinic, Cape Town, Western Cape